CLINICAL TRIAL: NCT01728714
Title: Prospective Study to Evaluate Impact of an Educational Programme About Diabetes, Comparing to Normal Clinical Practice, on Treatment Compliance and Disease Control of People With Type 2 Diabetes Followed in Primary Care Units in Portugal
Brief Title: Better Diabetes Control, Quality - Educate to Achieve Compliance.
Acronym: MINERVA
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-CPO-XXX-2012/1; CV/No drug/NIS-CPO-XXX-2012/1 (Other: CTT)
Record Dates: First submitted 2012-11-14; First posted 2012-11-20 (Estimated); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Diabetes Type 2
Keywords: Diabetes; compliance
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Patient Compliance

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Adults over 18 years old: Adults over 18 years old, with type 2 diabetes, HbA1c <= 8,5%, treated with oral antidiabetics at least for 6 months submitted to an educational programme during 1 year
- Adults with HbA1c <= 8,5%: Adults over 18 years old, with type 2 diabetes, HbA1c <= 8,5%, treated with oral antidiabetics at least for 6 months followed according to normal clinical practice during 1 year

SUMMARY:
Prospective study to evaluate the impact of an educational programme about diabetes, comparing to normal clinical practice, on treatment compliance and disease control of people with type 2 diabetes followed in the primary care units in Portugal

DETAILED DESCRIPTION:
Prospective study to evaluate the impact of an educational programme about diabetes focusing on treatment compliance, exercise and nutrition, comparing to normal clinical practice, on treatment compliance and disease control of people with type 2 diabetes followed in the primary care units in Portugal.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with type 2 diabetes
* HbA1c <= 8,5%
* Treated with oral antidiabetics for at least 6 months

Exclusion Criteria:

- Treatment with insulin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary care setting patients
Sampling Method: Probability Sample
Enrollment: 227 (Actual)
Dates: Start 2014-05-19 (Actual); Primary Completion 2018-12-05 (Actual); Study Completion 2018-12-05 (Actual)

PRIMARY OUTCOMES:
Number of people with type 2 diabetes treated with oral antidiabetics assessed as compliant with treatment after 1 year educational programme on diabetes, compared with normal clinical practice. | 1 year

SECONDARY OUTCOMES:
Number of people with type 2 diabetes treated with oral antidiabetics assessed as compliant with diet and physical exercise after 1 year educational programme on diabetes, compared with normal clinical practice. | 1 year
Number of people with type 2 diabetes treated with oral antidiabetics assessed as compliant with treatment with oral antidiabetics;after 1 year educational programme on diabetes, compared with normal clinical practice. | 1 year
Measure impact on quality of life, perceived by the patient, following 1 year educational programme on diabetes, compared with normal clinical practice. | 1 year
Measure the impact of compliance with treatment on glucose control following 1 year educational programme on diabetes, compared with normal clinical practice. | 1 year
Measure level of satisfaction of the patient with treatment and medical care following 1 year educational programme on diabetes, compared with normal clinical practice. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Cláudia Antão, Principal Investigator — Research Site 01; Pedro Carriço, Principal Investigator — Research site 02; Carla Gouveia, Principal Investigator — Research site 03; Jorge Vinagre, Principal Investigator — Research site 04
Locations (5):
- Portugal (5):
  - Research Site, Almada
  - Research Site, Espinho
  - Research Site, Loures
  - Research Site, Oeiras
  - Research Site, Santo Antonio Dos Cavaleiros

REFERENCES:
- See also: Abstract — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=NIS-CPO-XXX-2012/1&attachmentIdentifier=c39c2620-b385-4a20-9394-7e2059443955&fileName=MINERVA_Abstract_final_2023Apr17.pdf&versionIdentifier=